CLINICAL TRIAL: NCT02040545
Title: Venopuncture-Free IVF: Can "Patient-friendly" Salivary Hormone Measurements Replace Serum Monitoring of IVF Patients?
Brief Title: Salivary Diagnostic Testing for IVF
Status: Completed | Type: Observational
Sponsor: Boston IVF (Other)
Responsible Party: Principal Investigator, Alison Zimon, Reproductive Endocrinologist, Boston IVF
Other Study IDs: 20092198
Record Dates: First submitted 2013-05-21; First posted 2014-01-20 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: Infertility; In Vitro Fertilization (IVF); Venopuncture-free treatment; Needle-free treatment
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infertility: Patients undergoing ovulation induction and controlled ovarian hyperstimulation at a participating infertility center

SUMMARY:
This study aims to determine the performance of a salivary hormone competitive immunoassay for monitoring patients during treatment for infertility.

DETAILED DESCRIPTION:
The goal of this study is to determine the performance of a salivary hormone competitive immunoassay for monitoring patient estrogen and progesterone levels during treatment for infertility using controlled ovarian stimulation (COH) and in vitro fertilization (IVF). Specifically, inter- and intra-assay precision, correlation with serum measurements (the gold-standard), and user satisfaction will be determined. Ultimately, the potential applicability and reliability of salivary steroid monitoring in IVF cycles will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing In Vitro Fertilization (IVF) at a participating infertility center

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing In Vitro Fertilization (IVF) at a participating infertility center
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2010-05-21 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Equivalence of Salivary Steroid Monitoring to Blood Based Monitoring | 1 month
  The potential applicability and reliability of salivary steroid monitoring during infertility treatment will be measured as a progression during a patient's IVF stimulation cycle. Concurrent saliva and blood draw measurements of Estradiol and Progesterone will be taken between 3-5 times during a 2-week monitoring period. Equivalence will be determined by the matched progression of Estradiol and progesterone levels (pg/ml) in the same patient at the concurrent times. Saliva Estradiol and Progesterone levels are of a magnitude of 100-200 less than serum based values and are converted using an algorithm to adjust to serum equivalence. Matched T-test will be used to test the hypothesis that the two methods are not statistically different.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Zimon, MD, Principal Investigator — Boston IVF
Locations (8):
- United States (8):
  - HRC Fertility, Pasadena, California
  - Reproductive Biology Associates, Atlanta, Georgia
  - Fertility Center of Illinois, Chicago, Illinois
  - Boston IVF, South Portland, Maine
  - Shady Grove Fertility Reproductive Science Center, Rockville, Maryland
  - Boston IVF, Quincy, Massachusetts
  - Boston IVF, Waltham, Massachusetts
  - Reproductive Medicine Associates of New York, LLP, New York, New York

IPD SHARING:
Plan to Share IPD: No